CLINICAL TRIAL: NCT04808102
Title: Randomized Controlled Trial to Evaluate the Effectiveness of a Serious Game Targeting Interpersonal Emotion Regulation in Early Adolescents
Brief Title: The Effectiveness of a Serious Game Targeting Interpersonal Emotion Regulation in Early Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karl Landsteiner University of Health Sciences (Other)
Collaborators: Ludwig Boltzmann Gesellschaft (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DOT2021P1
Record Dates: First submitted 2021-03-16; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-02

CONDITIONS: Interpersonal Relations
Keywords: interpersonal emotion regulation; serious games; early adolescence

STUDY DESIGN:
Intervention Model Description: This trial is a RCT with an experimental and a control group, with participants being individually allocated to either of the groups. The allocation ratio is 50:50. This RCT adopts a pre-post-test strategy with the between-participant factor "group" and the within-participant factor "time".
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigator and trial participants will be blinded throughout the study due to the automised randomization process via the online server SosciSurvey. Statistical analysis will be executed by generating a number for each group, with its affiliation unknown to the analyst.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IER serious game (Experimental): A serious game training interpersonal emotion regulation strategies.
  Interventions: Device: IER AG
- control game (Sham Comparator): A control puzzle game without psychoeducational content.
  Interventions: Device: BubbleShooter

INTERVENTIONS:
Device: IER AG — The game is a web-based single-player adventure game with 3 levels created with the RPG Maker MV. Playtime is approximately 3 hours.
  Arms: IER serious game
Device: BubbleShooter — A free-to-play arcade browser puzzle game called BubbleShooter.
  Arms: control game

SUMMARY:
Background: Adaptive interpersonal emotion regulation (iER) is a vital tool for positive relations. During early adolescence, peer relations become increasingly important, making this age group a relevant target group for interventions promoting positive interactions with each other, yet no evidence-based intervention exists for early adolescents specifically.

Methods: This randomized controlled trial (RCT) aims to test effectiveness and feasibility of a serious game training iER skills in early adolescents by comparing outcomes with a control group playing a game without psychoeducational content in a pre- and post-test design. German- and English-speaking early adolescents (10-14 years) are eligible for participation. IER skills improvement assessed by a vignette task is the primary outcome variable and will be analysed with a chi-square test. Feasibility and acceptability and variables such as emotional competence, personal emotion regulation, gender, and sex will be assessed by questionnaires.

Discussion: This RCT will test whether playing serious game about iER strategies will result in an improvement of iER skills and whether the game is feasible and acceptable for early adolescents with the ultimate aim to implement the game in school classes and help early adolescents achieve positive peer relationships.

ELIGIBILITY:
Inclusion Criteria:

* Between 10 and 14 years old
* Willing and able to provide written parental consent
* Willing and able to participate in filling out pre- and post-test online questionnaires, and playing a web-based game
* Able to read and understand German or English
* Access to a device with internet (computer, mobile phone, tablet)

Exclusion Criteria:

-

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Interpersonal emotion regulation | The follow-up will be approximately 5 days after baseline measures.
  change of iER strategies participants can think of from pre (baseline)- to post-intervention, i.e. if the percentage of participants who improve their knowledge about possible iER strategies is higher in the experimental group compared to the control group. This is done via a vignette-task.

CONTACTS AND LOCATIONS:
Overall Officials: Beate Schrank, Study Director — Karl Landsteiner University of Health Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mittmann G, Zehetmayer S, Schrank B. Study protocol for a randomised controlled trial to evaluate the effectiveness of a serious game targeting interpersonal emotion regulation in early adolescents. Trials. 2021 Oct 25;22(1):741. doi: 10.1186/s13063-021-05706-7. PMID 34696816